CLINICAL TRIAL: NCT06752772
Title: WeArable teChnology daTa driVen digitAl healTh cOachINg (ACTIVATION)- A Mixed-methods Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandra Hospital (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DSRB2023/00276
Record Dates: First submitted 2024-07-25; First posted 2024-12-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Elevated Blood Pressure; Hypertension; Overweight/Obesity; Type 2 Diabetes Mellitus (T2DM); Hyperlipidemia; Prediabetes
Keywords: Digital Health Intervention; Health Coaching; Personalisation; Nudging; Wearables
MeSH Terms: conditions — Hypertension; Overweight; Obesity; Diabetes Mellitus, Type 2; Hyperlipidemias; Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Smart Watch only (Active Comparator): Participants will need to undergo HbA1c and lipid blood tests to determine if they have pre-diabetes, diabetes, or hyperlipidemia if they lack recent blood results (within 3 months prior to enrolment) for blood glucose and/or lipid levels.
  Participants assigned to Group 1 are required to fill out questionnaires covering aspects such as sociodemographic, lifestyle, medical condition, healthcare utilisation, quality of life, self-efficacy, distress and personality measures at study baseline, as well as at 3-, 6-, 9-, and 12-months following study enrolment.
  Participants will be issued a Fitbit Smartwatch and are required to wear the smart watch for at least 8 hours a day for a total duration of 6 months. Participants are encouraged to continue their normal daily activities while wearing the smart watch.
  Interventions: Device: Smart watch
- Group 2: Smart watch + dashboard with nudging system (Active Comparator): Participants will need to undergo HbA1c and lipid blood tests to determine if they have pre-diabetes, diabetes, or hyperlipidemia if they lack recent blood results (within 3 months prior to enrolment) for blood glucose and/or lipid levels.
  Participants assigned to Group 2 are required to fill out questionnaires covering aspects such as sociodemographic, lifestyle, medical condition, healthcare utilisation, quality of life, self-efficacy, distress and personality measures at study baseline, as well as at 3-, 6-, 9-, and 12-months following study enrolment.
  Participants will be issued a Fitbit Smartwatch and are required to wear the smart watch for at least 8 hours a day for a total duration of 6 months. Participants are encouraged to continue their normal daily activities while wearing the smart watch.
  Interventions: Device: Smart watch; Behavioral: Dashboard with nudging system
- Group 3: Smart watch + dashboard with nudging system + Digital Health Coach (DHC) (Experimental): Participants will need to undergo HbA1c and lipid blood tests to determine if they have pre-diabetes, diabetes, or hyperlipidemia if they lack recent blood results (within 3 months prior to enrolment) for blood glucose and/or lipid levels.
  Participants assigned to Group 3 are required to fill out questionnaires covering aspects such as sociodemographic, lifestyle, medical condition, healthcare utilisation, quality of life, self-efficacy, distress and personality measures at study baseline, as well as at 3-, 6-, 9-, and 12-months following study enrolment.
  Participants will be issued a Fitbit Smartwatch and are required to wear the smart watch for at least 8 hours a day for a total duration of 6 months. Participants will be assigned to a DHC and the DHC will be providing you with remote health coaching assistance for a duration of 6 months.
  Participants are encouraged continue their normal daily activities while wearing the smart watch.
  Interventions: Device: Smart watch; Behavioral: Dashboard with nudging system; Device: Digital Health Coach (DHC)

INTERVENTIONS:
Device: Smart watch — Participants are required to wear the study issued smart watch for at least 8 hours a day during the intervention period and are encouraged to wear it beyond the study intervention period.
Behavioral: Dashboard with nudging system — Nudges will be sent to participants' smart watch/mobile application with messages that are designed to motivate them to lead a healthy lifestyle.
  Arms: Group 2: Smart watch + dashboard with nudging system; Group 3: Smart watch + dashboard with nudging system + Digital Health Coach (DHC)
Device: Digital Health Coach (DHC) — Participants will be assigned to a DHC and the DHC will be providing them with remote health coaching assistance for a duration of 6 months, upon successful enrolment.
  Arms: Group 3: Smart watch + dashboard with nudging system + Digital Health Coach (DHC)

SUMMARY:
Public health priorities have shifted towards disease prevention, emphasising health promotion and lifestyle interventions to reduce disease burden. Despite global efforts, the prevalence of chronic diseases remains high, with lifestyle factors such as alcohol consumption, diet, smoking, obesity, and sedentary behaviour playing significant roles. In Singapore, suboptimal lifestyle behaviours are common, contributing to a high incidence of chronic conditions. Metabolic syndrome (MetS), linked to obesity, poses a growing societal burden due to its association with cardiovascular risks. Disparities exist in the delivery of lifestyle interventions among healthcare providers (HCPs), with many patients receiving inadequate guidance. Digital health coaching, incorporating wearable technology, offers promising solutions to bridge these gaps, providing personalised, real-time support and feedback to improve lifestyle behaviours and prevent disease progression. Challenges such as time constraints, lack of feedback, and limited support can be addressed through remote monitoring and tailored interventions, making scalable population-level interventions feasible.

ELIGIBILITY:
Inclusion Criteria:

* 21-75 years old
* Patients who are at risk of any of the following:

  1. Elevated blood pressure
  2. Overweight (BMI>=23kg/m2)
  3. Pre-diabetes, OR
* Patients who have one or more of the following (HOLD) conditions:

  1. Hypertension
  2. Obesity (BMI>=27.5kg/m2)
  3. HyperLipidemia
  4. Type 2 Diabetes Mellitus
* Patients who own a smartphone
* Patients who are willing to wear a smartwatch during the intervention period.

Exclusion Criteria:

* Patients who have a medical condition that prevented participation in physical activity
* Patients who have current diagnosis or history of eating disorder, depression
* Patients who are currently pregnant or planning to become pregnant in the next 6 months
* Patients who are currently participating in a weight loss programme (commercial, medically supervised, or research study)
* Patients who are on weight loss medications (over-the-counter or prescription)
* Patients who are not mentally-, physically- or technologically-capable
* Patients who is unable to provide informed consent.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Changes in physical activity level | Baseline, 6- and 12-month post study enrolment
  Change in physical activity level will be measured using the International Physical Activity Questionnaire Short Form (IPAQ-SF) scale at baseline, 6- and 12-month post study enrolment. Higher score indicates a higher level of physical activity.

SECONDARY OUTCOMES:
Engagement and sustainability | Baseline, 3- , 6-, 9-, and 12-month post study enrolment
  Duration of wearables wear time will be assessed throughout the study.
Acceptability of the study | 6-, 9- and 12-month post study enrolment
  In-depth qualitative interviews will be conducted to assess acceptability of the study.
Satisfaction towards the intervention provided | 6-month post study enrolment
  Satisfaction will be measured through Client Satisfaction Questionnaire (CSQ-8) for Group 3 participants. CSQ-8 uses a 4-point Likert scale, with higher score indicating greater satisfaction.
Lifestyle changes (Diet) | Baseline, 6-, and 12-month post enrolment
  Changes in diet intake will be measured through Healthy Eating Assessment (HEA) scale. Health Benefit score is calculated, and a higher score indicates that participants are in a possible healthier benefit zone.
Lifestyle changes (Smoking Cessation) | Baseline, 6-, and 12-month post enrolment
  Changes in smoking behaviour will be measured through Cigarette Dependence Scale (CDS-12). Higher score indicates a greater level of possible cigarette dependence.
Lifestyle changes (Alcohol Cessation) | Baseline, 6-, and 12-month post enrolment
  Changes in alcohol consumption will be measured through Alcohol User Disorders Identification Test (AUDIT). Higher score indicates a greater level of possible alcohol dependence.
Self-efficacy | Baseline, 6-, and 12-month post enrolment
  Self-efficacy will be measured through General Self-Efficacy (GSE) Scale. Higher score indicates a greater level of self-efficacy.
Quality of Life | Baseline, 6-, and 12-month post enrolment
  Changes in quality of life will be measured through EuroQol 5-Dimension 5-Level Health Questionnaire (EQ-5D-5L). Index scores closer to 1 indicates a better possible health state; a higher EQ-VAS score closer to 100 indicates a better possible health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No